CLINICAL TRIAL: NCT01652105
Title: Comparison of Preoperative Diets Before Bariatric Surgery: a Randomized Controlled Trial
Brief Title: Randomized Trial of Preoperative Diets Before Bariatric Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Lievensberg Ziekenhuis (Other)
Responsible Party: Principal Investigator, R. Schouten, MD, PhD, Lievensberg Ziekenhuis
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: rubenschouten1
Record Dates: First submitted 2012-07-25; First posted 2012-07-27 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-08

CONDITIONS: Morbid Obesity; Bariatric Surgery; Gastric Bypass
Keywords: Gastric bypass; Preoperative diet; Prodimed
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diet (Experimental): New developed diet
  Interventions: Dietary Supplement: Standard diet versus standard VLCD (Prodimed)
- Prodimed (Active Comparator): Standard VLCD
  Interventions: Dietary Supplement: Standard diet versus standard VLCD (Prodimed)

INTERVENTIONS:
Dietary Supplement: Standard diet versus standard VLCD (Prodimed)

SUMMARY:
Randomized clinical trial of two preoperative diets before bariatric surgery (gastric bypass)comparing standard diet and Prodimed (VLCD) in 100 morbidly obese patients selected for a gastric bypass procedure

DETAILED DESCRIPTION:
Morbid obesity, defined as a body mass index (BMI) of > 40 kg/m² or > 35 kg/m² with obesity-related comorbidities, is a rapidly growing problem in the western society. In the United States, about 6 million people currently have a BMI of > 40 kg/m² and another 10 million people have a BMI of > 35 kg/m² with comorbidities. Worldwide, the incidence of morbid obesity has doubled and about 300 million people are now obese. In the Netherlands the prevalence is less disturbing but the incidence of morbid obesity is rising progressively to 1.5% of the total population. At this moment surgical therapy is the only treatment option for these patients that results in sufficient long-term weight loss. Non-surgical approaches, like low energy diets and behavior modification, are not successful in the long-term with respect to maintaining weight loss and decreasing obesity-related comorbidities.

In order to increase weight loss and minimize complications a preoperative diet before bariatric has been advocated. However, the usual VLCD's are poorly tolerated by patients. In this study we aim to compare two preoperative diets in order to find the most suitable for this patient population.

ELIGIBILITY:
Inclusion Criteria:

* morbid obesity according to IFSO criteria

Exclusion Criteria:

* previous bariatric or gastric surgery
* severe psychiatric disorders

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-09; Primary Completion 2013-03 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Preoperative weight loss before bariatric surgery | 2 weeks
  Weight loss in kg before operation

SECONDARY OUTCOMES:
- operation time - blood loss - difficulty of procedure - short term complications - acceptance of diets according to patients | 2 weeks
  Measured by VAS, diet books and questionnaires

CONTACTS AND LOCATIONS:
Locations (1):
- Bariatric Centre Lievensberg hospital, Bergen op Zoom, Netherlands